CLINICAL TRIAL: NCT05581862
Title: Effect Of Meal Frequency On Weight Loss And Body Composition Of Obese And Overweight Women Having Medical Nutrition Therapy
Brief Title: Effect Of Meal Frequency On Weight Loss And Body Composition Of Obese And Overweight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/21-03
Record Dates: First submitted 2022-10-05; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Overweight and Obesity
Keywords: Meal Frequency; body composition; BMI; waist circumference
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 Meals+3 Snacks (Experimental): This group was followed up for 3 months with an energy restricted weight loss plan composed of 3 main meals and 3 snacks
  Interventions: Behavioral: 3 meals+3 snacks
- 3 Meals (Experimental): This group was followed up for 3 months with an energy restricted weight loss plan composed of 3 main meals
  Interventions: Behavioral: 3 meals

INTERVENTIONS:
Behavioral: 3 meals+3 snacks — All of the 20 subjects consumed an energy restricted weight loos plan with 3 main meals and 3 snacks for 3 months
  Arms: 3 Meals+3 Snacks
Behavioral: 3 meals — All of the 20 subjects consumed an energy restricted weight loos plan with 3 main meals for 3 months
  Arms: 3 Meals

SUMMARY:
Studies showing the relationship between meal frequency, weight loss and anthropometric measurements are contradictory. This study is planned and conducted to observe the effects of meal frequency (3 meals+3 snacks vs 3 meals) on weight loss, anthropometric measurements and body composition with 3-month energy restricted Medical Nutrition Therapy program in 19-64 years old women with a BMI ≥ 27 kg/m2.

DETAILED DESCRIPTION:
The study was conducted with 40 female volunteers between the ages of 19-64 years, with a Body Mass Index (BMI) ≥27. Energy restricted individualized weight loss programs were applied with different meal frequencies (3 meals+3 snacks/day vs 3 meals/day) in a 3 month follow up period. 20 participants were randomized in 3 meals+3 snacks and 20 participants were randomized in 3 meals group. Food consumption was questioned, and anthropometric measurements and body composition were measured before the study and repeated each week till the end of the study. Three day food records (2 week days and 1 weekend day) taken before the intervention were evaluated and five hundred calorie was subtracted from the average energy calculated form the food records to determine the energy of the weight loss plans . Breakfast, lunch and dinner are planned as main meals and the beverages and/or food eaten between main meals were planned as snacks (50-200 kcal). For both of the groups dietary weight loss program was planned by the same dietitian. Macronutrient composition of the weight loss plan was designed according to the recommendations of the Turkish Dietary Guidelines as 45-60 % carbohydrate, 10-20 % protein and 20-35 % fat for both of the groups.

ELIGIBILITY:
Inclusion Criteria:

* 19-64 years old Women,
* Healthy subjects with no chronic diseases,
* Subjects who were not taking any drug or dietary supplements,
* Subjects who have not made any changes in their physical activity or eating habits for weight loss in the last 6 months,
* Subjects with a BMI ≥ 27 kg/m2

Exclusion Criteria:

* Failure to meet the criteria for inclusion

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in BMI (kg/m2) | 3 months
  Both of the groups had a significant change in BMI, but there was no difference among the groups
Change in Waist circumference (cm) | 3 months
  Both of the groups had a significant change in waist circumference, but there was no difference among the groups
Change in total body fat (kg) | 3 months
  Both of the groups had a significant change in total body fat however the rate of change in total body fat was significantly higher in 3 meals+3snacks group
Change in body fat percentage (%) | 3 months
  Both of the groups had a significant change in body fat percentage however the rate of change in body fat percentage was significantly higher in 3 meals+3snacks group
Change in fat free mass percentage (%) | 3 months
  Both of the groups had a significant change in fat free mass percentage, however the rate of change was significantly higher in 3 meals+3 snacks group

CONTACTS AND LOCATIONS:
Overall Officials: Müjgan Öztürk, PhD, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otuken Koroglu Y, Ozturk M. Meal Frequency Does Not Affect Weight Loss in Overweight/Obese Women but Affects the Body Composition: A Randomized Controlled Trial. J Am Nutr Assoc. 2024 Aug;43(6):489-497. doi: 10.1080/27697061.2024.2316636. Epub 2024 Feb 13. PMID 38349951